CLINICAL TRIAL: NCT05933421
Title: A Single Center Retrospective Cohort Study of Auto-intoxicated Patients Admitted to the ICU: Descriptive Analysis
Brief Title: A Single Center Retrospective Cohort Study of Auto-intoxicated Patients Admitted to the ICU
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Dr, PhD, Jessa Hospital
Other Study IDs: f/2023/041
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Intoxication, Depth
MeSH Terms: conditions — Inert Gas Narcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intentional poisoning is a relevant public health issue responsible for a considerable number of cases of morbidity and mortality worldwide. There are no concrete numbers/investigations of these patients admitted to the ICU at our hospital, with limited insight on their characteristics and outcome.

It is expected that this population of patients is an important burden for the ICU. It can be important to shed a light on prevalence and ratio of intoxicated patients admitted to the ICU in our center.

Furthermore, during the covid-pandemic, we could expect an increase in self-poisoning prevalence due to social restrictions, more limited access to (mental) health care, etc…

DETAILED DESCRIPTION:
Aim The aims of this study are to quantify the ratio of intensive care admissions attributable to self-poisoning in our hospital, to examine characteristics and outcome of these patients, yearly trends and impact of the covid-pandemic on these variables.

Design A single center retrospective cohort study analysis of patients with self-poisoning admitted to ICU of the Jessa Hospital Hasselt Belgium over a period of 6 years (2017-2022).

Sample size

All patients diagnosed with self-poisoning admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022 were included in the study. This were 377 patients.

Study population

Inclusion and exclusion criteria:

All patients (>14 years of age) diagnosed with self-poisoning and admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022 were included in the study.

Patient admitted for tentamen suicide but not due to intoxication were excluded as well as patients with no medical records in the Jessa hospital.

Primary Outcome The prevalence of auto-intoxicated patients admitted to the ICU together with the mortality rate on the ICU.

Secondary Outcome measurements

Secondary outcome measurement are the ICU and hospital length of stay, ratio of auto-intoxicated patients to all patients admitted at ICU, types of drugs ingested, number of drugs involved, cause of admission, yearly trends and impact of covid-pandemic.

Statistical analysis Data will be presented as mean values +/-SD, numbers(n), and percentages(%) or median (25%, 75% percentile) in case of non-parametric data. Categorical variables are presented as frequencies (%) and groups were compared using Chi-square or Fisher's exact test.

Differences between patients change will be analyzed using the Student t test for continuous outcomes or, in case of non-parametric data, the Mann-Whitney U test. Univariate and multivariate logistic regression models will be used in order to predict mortality. P values <0.05 will be considered statistically significant.

Additional data collection:

Additional collected parameters are listed below and are collected as a standard-of-care in our hospital:

* Demographics: i.e age, gender, BMI
* DNR-code
* Admission route
* Patient state and symptoms: i.e vital signs, GCS, …
* Comorbidities: i.e smoking, obesity, hypertension, diabetes, cardiovascular disease, respiratory disease, malignancies, renal failure, liver failure, neurological conditions, mental state and disease
* Technical investigation results: i.e Laboratory results, ECG, radiological findings, etc…
* Complications: i.e shock, heart failure, sepsis, stroke, etc…
* Ventilation: method, PEEP, FiO2, P/F ratio,…
* Management: i.e antidote, supportive, mechanical ventilation, dialysis, observation,

ELIGIBILITY:
Inclusion Criteria:

All patients (>14 years of age) diagnosed with self-poisoning and admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022 were included in the study.

Exclusion Criteria:

Patient admitted for tentamen suicide but not due to intoxication were excluded as well as patients with no medical records in the Jessa hospital.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (>14 years of age) diagnosed with self-poisoning and admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of mortality | patient admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022
  The prevalence of auto-intoxicated patients admitted to the ICU together with the mortality rate on the ICU.

SECONDARY OUTCOMES:
ICU length of stay | patients admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022
  Length of stay in the ICU
hospital length of stay | patients admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022
  Length of stay in the hospital
Relative number of auto-intoxicated patients at ICU | patients admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022
  ratio of auto-intoxicated patients to all patients admitted at ICU,
Type | patients admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022
  type of drugs ingested by patients admitted to ICU
number of drugs or medication | patients admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022
  number of drugs or medication ingested by patients admitted to ICU
Cause | patients admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022
  cause of admission to ICU: emotional, relational, somatic, psychological, financial, workrelated, recreative, other or unknown
Impact of COVID-19 pandemic | patients admitted to the ICU of the Jessa hospital between 01/01/2017 and 31/12/2022
  the impact of the COVID-19 pandemic on the number of auto-intoxicated patients admitted to ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No